CLINICAL TRIAL: NCT03109743
Title: Development and Testing of a Group Clinical Visit Adherence Intervention for HIV+ Women of Color
Brief Title: Group Clinical Visit Adherence Intervention for HIV+ Women of Color
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The funding for the study was relinquished and so study terminated early.
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Albert Einstein College of Medicine (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Oni Blackstock, Assistant Professor, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016-7257; K23MH102129 (NIH)
Record Dates: First submitted 2017-04-06; First posted 2017-04-12 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Adherence, Patient; HIV/AIDS; Group Meetings
Keywords: HIV treatment; Adherence Group Treatment
MeSH Terms: conditions — Patient Compliance; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: The investigators pilot test efficacy of Sisters-GPS intervention in improving ARV adherence by randomizing 60 HIV+ women of color with suboptimal ARV adherence and detectable HIV viral loads (VL) to Sisters-GPS, group clinical visits, or to an appointment with an adherence counselor. The investigators will collect data from interviews, pill counts, medical and pharmacy records, and blood samples. The study's primary outcome will be ARV adherence assessed by pill count at 8 weeks; secondary outcome will be change in HIV VL from baseline to 8 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sisters-GPS: Group Clinical Visits (Experimental): Those randomized to the Sisters-GPS arm will be expected to attend a total of seven group clinical visits, once a week for ~1.5 hours. Groups visits will include education, self-management skills development, and a clinical assessment by a medical provider with a focus on HIV treatment and adherence. Additionally, Sisters-GPS participants will be encouraged to participate in a private social media site specifically designed for the study, where participants will be able communicate with one another and with research staff. Group size will be 8-10 participants.
  Interventions: Behavioral: Sisters-GPS: Group Clinical Visits
- Control: One-on-one Adherence Counseling (Active Comparator): Those randomized to the control condition will receive an appointment with a HIV treatment adherence counselor and will be expected to attend a minimum of three adherence counseling visits. .
  Interventions: Behavioral: Control: One-on-one Adherence Counseling

INTERVENTIONS:
Behavioral: Sisters-GPS: Group Clinical Visits — Sisters-GPS will be involve group clinical visits where by the same group participants with meet with a clinician and behaviorist to receive education, self-management skills development, and clinical assessment over the seven weekly group visits. The content will focus specifically on HIV medications and medication adherence. Additionally, the intervention will involve a private social media website where participants will be able to engage with one another between group clinical visits. Participants will receive food and a roundtrip Metrocard at each group clinical visit.
  Arms: Sisters-GPS: Group Clinical Visits
Behavioral: Control: One-on-one Adherence Counseling — For participants in the control arm, the counselor will provide standard-of-care adherence counseling, which includes education about ARVs and the importance of adherence, and addressing non-adherence including assessment of psychosocial barriers to adherence. For visits to the adherence counselor, participants will receive round-trip MetroCards as per clinic policy. Control arm participants will be expected to attend a minimum of three visits with the adherence counselor.
  Arms: Control: One-on-one Adherence Counseling

SUMMARY:
The investigators will conduct a pilot randomized controlled trial (RCT) of Sisters-GPS with HIV-positive women of color with suboptimal ARV adherence and detectable HIV viral loads (VL). Participants will be randomized to Sisters-GPS (intervention involving weekly group clinical visits for seven weeks plus social media website) or appointment with an adherence counselor (a minimum of 3 visits) (control condition). Data sources will include interviews, medical and pharmacy records, and blood samples. The primary outcome will be ARV adherence at the completion of the intervention assessed via pill count. The secondary outcome will be HIV VL suppression.

DETAILED DESCRIPTION:
African American and Latina women comprise about 80% of the approximately 300,000 HIV-positive women in the United States. HIV/AIDS is one of the leading causes of death among African American and Latina women age 20 to 55 years. HIV-positive women of color are disproportionately impacted by poverty and other factors such as substance abuse and mental illness which increase vulnerability to HIV and risk of poor health outcomes (e.g., progression to AIDS and death).

The stages of HIV treatment cascade include linkage to and retention in HIV care, antiretroviral (ARV) utilization, and viral suppression. While all of these stages are important, what has ultimately lengthened life expectancy among HIV-positive persons has been achieving long-term viral suppression by optimizing ARV adherence. Suboptimal ARV adherence is associated with increased risk of progression to AIDS, mortality, and the development of ARV resistance. Recent studies indicate that significant racial and ethnic disparities in ARV adherence persist, with African Americans and Latinos having lower levels of adherence than whites. This disparity is also reflected among HIV+ women, with women of color, and in particular African American women, having significantly lower rates of ARV adherence than white women.

Peer-based health interventions have been shown to affect behavior and improve patient outcomes. For HIV-positive persons, receiving care within a group of peers is associated with decreased levels of shame, HIV-related stigma, and risk behaviors, and increased levels of perceived social support. A group-based approach to care involving peers may be especially important for HIV-positive women of color as HIV-positive women of color may lack positive social support. Consequently, the peer-group dynamic may help not only to normalize living with HIV and provide social support but also to motivate healthy behaviors such as ARV adherence.

Group clinical visits, in which the same group of patients who share a common medical condition receives care simultaneously from a health care provider over time, is a model of care that seeks to take advantage of the peer-group dynamic. This model often includes a clinical assessment, education, and self-management skills development, all in the group setting. It has been utilized in the care of patients with chronic conditions such as diabetes mellitus and Hepatitis C infection and improves health outcomes. Therefore, guided by an enhanced version of the Social Learning Theory, which posits that people learn not only from their own experiences but from the experiences and actions of others, the investigators will tailor the group clinical visit model to a model of group HIV treatment focused on optimizing ARV adherence.

Use of social media, whereby people interact by creating, sharing, and exchanging content using internet-based technologies, transcends race/ethnicity and socioeconomic status. Within the arena of health care, its use is becoming increasingly popular. For example, social media is used by persons who may have a common medical condition, such as HIV, to communicate about coping with the disease or taking medications. Among HIV-positive persons, social media may be used to enhance communication and social support; hence, the investigators have incorporated social media as a component of Sisters-GPS.

To begin to address disparities in ARV adherence and the limitations of current interventions, the investigators will test Sisters-GPS, an intervention for HIV-positive women of color with suboptimal ARV adherence that the investigators have developed. Sisters-GPS is an intervention adapted from the group clinical visit and which incorporated social media. If proven effective, this intervention has the potential to be a model of health care delivery for HIV care and treatment, more generally, and can be disseminated to diverse clinical settings.

ELIGIBILITY:
Inclusion criteria:

1. HIV-positive
2. Cis gender women (assigned female sex at birth and current identifies as female)
3. ≥ 18 years old
4. English proficiency
5. At least one visit to community health center where received HIV primary care within the last 12 months
6. Self-reported ARV adherence <100% in the previous 30 days
7. Most recent HIV viral load in last 12 months detectable
8. Prescribed HIV medications for at least 16 weeks prior to detectable HIV viral load
9. Currently prescribed HIV medications (i.e., current active HIV medication prescription in electronic medical record or pharmacy)
10. Able to attend most/all group visits

Exclusion Criteria:

1. Untreated severe mental illness including major depressive disorder, bipolar disorder, schizophrenia, psychosis, or current suicidal ideation.
2. Acute intoxication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Individual assigned female sex at birth and who currently identify as female.
Enrollment: 15 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2017-12-07 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
Antiretroviral Therapy (ARV) adherence | 8 weeks
  Pill count, self-report

SECONDARY OUTCOMES:
Change in HIV viral load | 8 weeks
  Change in HIV viral load from baseline to 8 weeks modeled as continuous variable
HIV Viral Load (VL) suppression | 8 weeks
  HIV VL used as a dichotomous measure (VL<40 copies/mL, yes/no)
Antiretroviral Therapy (ARV) adherence | 4 weeks
  Pill count, self-report
Antiretroviral Therapy (ARV) adherence | 20 weeks
  Pill count, self-report
HIV Viral Load (VL) suppression | 20 weeks
  HIV VL used as a dichotomous measure (VL<40 copies/mL, yes/no)
Change in HIV viral load | 20 weeks
  Change in HIV viral load from baseline to 8 weeks modeled as continuous variable

OTHER OUTCOMES:
ARV beliefs and attitudes | at baseline, 4 weeks, 8 weeks, 20 weeks
  Measure using an ARV beliefs and attitudes questionnaire
ARV Knowledge | at baseline, 4 weeks, 8 weeks, 20 weeks
  Measure using a HIV Treatment Knowledge Scale
Medication side effects | at baseline, 4 weeks, 8 weeks, 20 weeks
  Measure using Treatment Satisfaction Questionnaire for Medication
Perceived self-efficacy | at baseline, 4 weeks, 8 weeks, 20 weeks
  Measure using an ARV adherence Self-Efficacy Scale
Perceived HIV-related stigma | at baseline, 4 weeks, 8 weeks, 20 weeks
  Measure using the HIV Stigma Scale
Perceived social support | at baseline, 4 weeks, 8 weeks, 20 weeks
  Measured using Scale of Perceived Social Support

CONTACTS AND LOCATIONS:
Overall Officials: Oni Blackstock, MD, MHS, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No